CLINICAL TRIAL: NCT07242963
Title: Registry Study of Children and Adults Patients With Relapsed, Refractory, or Progressive Sonic Hedgehog Medulloblastoma Harboring U1 Mutation
Brief Title: Relapsed and Progressive Sonic Hedgehog Medulloblastoma With U1 Mutation Registry Study
Status: Recruiting | Type: Observational
Sponsor: Mohammad H. Abu Arja (Other)
Collaborators: Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Mohammad H. Abu Arja, Instructor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: H-56521
Record Dates: First submitted 2025-11-07; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Medulloblastoma Recurrent; Medulloblastoma, Childhood, Recurrent; Medulloblastoma, SHH-activated and TP53 Mutant; Medulloblastoma, SHH-activated and TP53 Wildtype
Keywords: SHH medulloblastoma; medulloblastoma; medulloblastoma Recurrent
MeSH Terms: conditions — Medulloblastoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor samples: Tumor samples will be obtained from the residual samples after tumor resection for clinically indicated reasons. Frozen tumor samples and/or formalin-fixed paraffin-embedded tumor (FFPE) samples will be collected whenever available.
  Buccal samples: Buccal swabs will be collected using self-collection kits. Buccal swab samples will be requested from the patients and biological parents (if enrolled).
  Blood and cerebrospinal fluid (CSF) samples: Blood samples will be obtained and included for whole genome sequencing and intron detection. For CSF, we will collect existing (leftover) samples for future studies. For research samples, the study requests that the research samples be collected when serum samples are collected for clinical reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients treated at registry institutions
- Group 2: Patients not treated at registry institutions
- Group 3: Biological parents of a subject participating in Group 1 or 2

SUMMARY:
The purpose of this study is to create a biobank for patients diagnosed with Sonic Hedgehog Medulloblastoma at Baylor College of Medicine/Texas Children's Cancer Center. A biobank is a facility that stores and manages biological samples (such as blood, tissue, or DNA) from individuals, along with detailed health information, for use in medical research to study diseases and develop new treatments. The investigators are requesting participants' permission to add their information and samples to this biobank.

Being in this research study is voluntary; it is the participant's choice. If the participant joins this study, they can still stop at any time.

If the participant decides to participate, the investigators will review the participant's clinical medical records, demographics, treatment history, family history, and imaging. The investigators will also collect biological samples from the participant and the biological parents' buccal swabs (optional).

The participation in this biobank will last about 5 years from the decision to participate.

Why am I being asked to participate? The participant or their child is invited to participate in this study if the participant or their tumor may have a U1 mutation. U1 mutation is associated with an error in the gene that splices the tumor DNA, leading to random splicing that may increase the tumor mutation burden and generate novel tumor neoantigens (targets). Studying the U1 mutation will enable the investigator to design more effective therapies and guide future treatments for patients with relapsed or refractory sonic hedgehog medulloblastoma, thereby improving their outcomes and quality of life. Moreover, the investigators aim to determine whether germline mutations inherited from parents may increase the risk of medulloblastoma in their offspring. The participant will receive no direct benefit from their participation in this study. However, participation in this study may help the investigators better understand SHH Medulloblastomas and benefit other patients in the future.

DETAILED DESCRIPTION:
This is a multicenter, retro- and prospective observational cohort registry study. The registry will collect prospective data on children and young adults between ≥3 and ≤50 years of age at diagnosis, who are diagnosed with relapsed, refractory, or progressive SHH medulloblastoma. Patients and their biological parents will be recruited for this study. In addition, retrospective data will be gathered on patients enrolled in the registry to understand prior therapies and treatment courses before enrollment.

The local principal investigators will identify patients diagnosed at registry institutions through their clinical meetings and databases.

Patients diagnosed at non-registry institutions can get information on the registry through various sources, including but not limited to:

Clinicaltrials.gov registry information Texas Children's Cancer Center website Other patients enrolled in the registry Advertising through scientific talks/posters via various consortia, meetings, and patient support groups

Radiology: imaging studies for patients enrolled and treated in Texas Children's Cancer Center/Baylor College of Medicine (BCM) will be saved in their electronic medical records and uploaded to the radiology PACS system as part of their regular clinical care. For patients enrolled from outside treating centers, imaging CDs will be requested and sent by the legal guardian/patient. Personal health information will be redacted. The investigators will assign each CD a unique research acquisition number linked to the study subject. The study subjects will be assigned a unique study identifier, and images will be uploaded by the Texas Children's Radiology Department to the PACS system for reading. Only study-designated personnel will be allowed to access the imaging, and all published data will be de-identified. CDs will be stored in a locked cabinet.

Subjects at non-registry sites will request their treating centers to release their medical records, send tissue samples previously collected (if available), and release radiological imaging to the registry site (BCM). Patients or legal guardians will sign release forms at their treating centers to allow them to send the requested medical records, imaging, and tissue materials to the registry site (BCM). The enrolled patient or legal guardian will request the treating non-registry center to compile and send all the data to the registry site (BCM)

Primary and correlative studies performed on tissue will include the following:

U1 Mutation RNA-sequencing U1 Mutation PCR Methylation Profiling Intron detection via whole genome sequencing Whole genome sequencing RNA sequencing Spatial genomics & transcriptomics Proteomics Patient-derived xenografts (PDX) and cell lines generation Tissue banking Biological parental buccal swabs for whole genome sequencing

Data Protection Subjects will be assigned a unique identifier. Subject identifiers (e.g., name, medical record number) will be redacted from all samples. Only the investigator and personnel designated by them will have access to information that matches the study's unique identifier with patient-identifying information. If subjects withdraw from the study, they (or a legal guardian) may request the destruction of any samples taken and not tested, and the investigator must document this in the site study records. Because the purpose of the exploratory aims of the study is to facilitate IRB-approved research to develop new knowledge about the biology of SHH medulloblastoma that can be used to benefit patients in the future and not to provide clinical information, no test results will be routinely returned to study subjects or their oncologists. However, in rare cases in which research studies performed using the samples identify results for which significant clinical relevance has been clearly established through publication in peer-reviewed scientific journals, such results may be returned to the subject and/or their treating oncologist (only if the subject has provided specific consent for this optional procedure at the time of study enrollment). It will be emphasized to enrolled subjects that these are research results and must be confirmed in a clinical or diagnostic laboratory for clinical purposes.

In order to speed up research on SHH medulloblastoma, enrolled subjects will be given the option to allow their genetic and/or clinical data to be collected and analyzed as part of IRB-approved research protocols using tissue bank samples to be submitted into scientific databases, such as those maintained by the National Institutes of Health. It's important to note that these databases are highly secure and can only be accessed by approved researchers, ensuring the confidentiality and privacy of the participants' data. Only de-identified genetic and/or clinical information would be released for the NIH databases with subject consent.

Data Quality Quality control procedures for this research registry include source data verification by randomly selecting 10% of registry subject records by comparing the paper case report form (CRF) and the electronic database record of those same data. Quality control procedures will be performed at least once every 12 months by the principal investigators or their designees. If errors are common, data will be checked entirely before the data analysis.

Sample Size The planned sample size of 100 participants was used to estimate achievable precision, defined as the half-width of the 95% confidence interval for the point estimate of each primary outcome measure.

U1 Mutation Status The proportion of participants who harbor the U1 mutation amongst all enrolled participants is assumed to be 50%. With a sample size of 100 participants, the 95% confidence interval for U1 mutation status would have a half-width of at most 9.8% from the observed proportion.

Feasibility Given the assumption that 50% of participants who have SHH MB harbor the U1 mutation, the investigators estimate that out of 100 enrolled participants, 50 participants will have the U1 mutation by PCR and 50 will not. Given a target value of 95% for sensitivity, specificity, PPV, NPV, and accuracy of RNASeq (new diagnostic test), the 95% confidence intervals for these estimates would have half-widths of 6.0% at most.

Statistical Analyses General Baseline demographic, disease, and treatment characteristics will be summarized with mean and standard deviation or median and interquartile range for continuous variables, and counts and percentages for categorical variables. All analyses will be carried out using SAS (version 9.4 or higher) and R statistical software (version 4.5.0 or higher).

Primary Analyses U1 Mutation Status U1 mutation status, as determined by PCR, will be summarized in the overall sample and within each SHH medulloblastoma subtype with counts and percentages, along with the corresponding 95% confidence intervals.

Feasibility Sensitivity, specificity, PPV, NPV, and accuracy of the new RNASeq diagnostic test will be estimated, utilizing PCR as the reference standard. Only complete cases will be utilized in the following estimations.

Sensitivity will be estimated as the proportion of true positives (i.e., those testing positive with both RNASeq and PCR) out of all positive PCR tests, while specificity will be estimated as the proportion of true negatives out of all negative PCR tests. Positive predictive value will be estimated as the proportion of true positives out of all positive RNASeq tests, while NPV will be estimated as the proportion of true negatives out of all negative RNASeq tests. Finally, accuracy will be estimated as the proportion of true positives and true negatives out of all tests completed.

Sensitivity, specificity, PPV, NPV, and accuracy will be described as percentages, along with the corresponding 95% confidence intervals. In the event that there is discordance between RNASeq and PCR, the PCR result will be considered the "correct" result and the RNASeq result will be categorized accordingly (i.e., false positive or false negative). Any discordance will be summarized descriptively.

Secondary Analyses:

Overall survival, defined as time from enrollment to death from any cause, and event-free survival (EFS), defined as time from enrollment to progression, relapse, diagnosis of secondary cancer, change in therapy, or death from any cause, will be summarized descriptively by U1 mutation status and SHH MB subtype. Both OS and EFS will utilize the Kaplan-Meier method to estimate counts, time-specific rates, corresponding 95%confidence intervals, and survival curves. Early withdrawals and those remaining alive and event-free at the end of the study will be censored at the time of last know status. Subgroup analysis Given the interest in immune checkpoint inhibitor therapy and its effect on survival, OS and EFS will also be summarized amongst patients who received immune checkpoint inhibitors after enrollment on the study, both overall and by U1 mutation status, as time from initiation of immune checkpoint inhibitor therapy to the previously defined events. This subgroup analysis will be summarized using the same survival methods outlined above.

Interim Analyses No interim analyses are planned, as this is an observational study not designed for hypothesis testing.

Safety Given that this is an observational cohort study, patient safety with respect to adverse events will not be assessed.

ELIGIBILITY:
Inclusion Criteria:

For Groups 1 and 2, subjects are eligible to be included in the study only if all of the following criteria are met:

* Age Patients must be ≥ 3 and ≤ 50 years of age at the time of initial diagnosis.
* Diagnosis Participants must have a diagnosis of SHH medulloblastoma by histologic or molecular criteria at the time of original diagnosis or relapse.
* Disease status The disease must be recurrent, refractory, or progressive following therapy, including radiotherapy and chemotherapy.
* Available tumor tissue sample for U1 testing Participants must have available tumor tissue samples to be tested for the U1 mutation.

For Group 3, biological parent(s) of a subject participating in Group 1 or 2 are eligible.

Exclusion Criteria:

Subjects not meeting the inclusion criteria will be excluded.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Group 1 - Patients diagnosed/treated at Texas Children's Hospital (TCH) or one of the participating registry institutions.
  Group 2 - Patients diagnosed at non-registry institutions (an institution not participating in the registry as a site with IRB approval with BCM/TCH as the coordinating center).
  Group 3 - Biological parents of patients in Group 1 or 2.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2035-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
To describe the incidence of the U1 mutation in SHH medulloblastoma subtypes and verify the feasibility of U1 testing. The primary outcome will be detecting the U1 mutation by polymerase chain reaction (PCR) testing or RNA sequencing (RNAseq). | Through study completion, an average of 2 years
  U1 mutation status, as determined by PCR, will be summarized in the overall sample and within each SHH medulloblastoma subtype with counts and percentages, along with the corresponding 95% confidence intervals. Feasibility Sensitivity, specificity, PPV, NPV, and accuracy of the new RNASeq diagnostic test will be estimated, utilizing PCR as the reference standard. Only complete cases will be utilized in the following estimations. Sensitivity will be estimated as the proportion of true positives out of all positive PCR tests while specificity will be estimated as the proportion of true negatives. Positive predictive value will be estimated as the proportion of true positives out of all positive RNASeq tests. NPV will be estimated as the proportion of true negatives out of all negative RNASeq tests. Finally, accuracy will be estimated as the proportion of true positives and true negatives out of all tests completed.

SECONDARY OUTCOMES:
To collect and compare the outcomes of the different treatment regimens utilized for pediatric and adult patients with recurrent, refractory, or progressive SHH medulloblastoma with and without U1 mutation. | Through study completion, an average of 2 years
  Overall survival (OS) and event-free survival (EFS) will be summarized descriptively by U1 mutation status and SHH MB subtype. Both OS and EFS will utilize the Kaplan-Meier method to estimate counts, time-specific rates, corresponding 95% confidence intervals, and survival curves. Early withdrawals and those remaining alive and event-free at the end of the study will be censored at the time of last know status. No interim analyses are planned, as this is an observational study not designed for hypothesis testing. Given that this is an observational cohort study, patient safety with respect to adverse events, will not be assessed.

OTHER OUTCOMES:
To facilitate somatic and germline tissue testing to understand the unique biology of these rare tumors. | Through study completion, an average of 3 years
  Whenever available, tumor tissue will be requested pre- and post-treatment with or without immune checkpoint inhibition to uncover alterations in tumor biology secondary to treatment. Correlative studies performed on tissue will include the following:
  Methylation Profiling Intron detection via whole genome sequencing Whole genome sequencing RNA sequencing Spatial genomics & transcriptomics Proteomics Patient derived xenografts (PDX) and cell lines generation Tissue banking Biological parental buccal swabs for whole genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Murali Chintagumpala, MD, Study Chair — Baylor College of Medicine; Michael D Taylor, MD, PhD, Study Chair — Baylor College of Medicine; Mohammad H Abu-Arja, MD, MSc, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable. This study is an observational cohort study and not an interventional trial.